CLINICAL TRIAL: NCT06111989
Title: To Drive or Not to Drive? A Machine Learning Data Analysis Approach Among Stroke Patients
Brief Title: Fitness to Drive Among Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Institute for Medical Rehabilitation, Hungary (Other Government)
Collaborators: Semmelweis University (Other)
Responsible Party: Sponsor
Other Study IDs: IV/649-1/2022/EKU
Record Dates: First submitted 2023-09-06; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Driving Impaired
Keywords: fitness to drive; neuropsychology; cognitive; machine learning
MeSH Terms: conditions — Stroke | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: Patients who suffered ischemic or hemorrhagic stroke.
  Interventions: Behavioral: Neuropsychological testing; Behavioral: On road test

INTERVENTIONS:
Behavioral: Neuropsychological testing — The neuropsychological assessment will involve paper and pencil tests, computerized tests (such as reaction time measurements) and a driving simulator.
Behavioral: On road test — The driving instructor will guide the participant on a standard route, and will evaluate the performance using standard criteria that will focus mainly on traffic safety.

SUMMARY:
The goal of this observational study is to learn more about who can continue driving a car after a stroke. The focus of this study is on the relationship between cognitive abilities and fitness-to-drive.

Participants will be asked to perform an extended neuropsychological testing and a real life on-road test, conducted by a professional driving instructor. Feedback will be given to the participants on request.

DETAILED DESCRIPTION:
The relationship between cognitive abilities and driving skills is really complex. This study aims to introduce novel data analysing methods that can be used by medical professionals to decide whether the stroke patient is able to operate a vehicle safely or not.

The neuropsychological assessment will involve paper and pencil tests, computerized tests (such as reaction time measurements) and a driving simulator. This part will be approximately 2 hours. Since the first part is really tiresome, the test driving will be on an other day. The driving instructor will guide the participant on a standard route, and will evaluate the performance using standard criteria that will focus mainly on traffic safety.

Who can participate in the study:

* Aged 65 or younger
* Holds a driving licence
* Had an ischemic or hemorrhagic stroke
* Has sufficient physical abilities to operate a car
* Does not have certain medical conditions such epilepsy

ELIGIBILITY:
Inclusion Criteria:

* 65 or younger
* ischemic or hemorrhagic stroke
* at least 6 months has passed after the stroke
* holds a valid driver's licence

Exclusion Criteria:

* visual impairments (eg. visual field loss, nystagmus or diplopia)
* epilepsy
* serious movement disorders (eg. hemiplegia) that hider operating a car
* limb ataxia
* aphasia types that affect comprehension
* serious psychiatrical disorders

Max Age: 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients of the National Institute for Medical Rehabilitation, Budapest, Hungary
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Driving test result | through study completion, an average of 2 years
  The driving instructor's classification (pass/fail)

CONTACTS AND LOCATIONS:
Overall Officials: Gábor Fazekas, MD, PhD, Principal Investigator — National Institute for Medical Rehabilitation, Hungary
Locations (1):
- National Institute for Medical Rehabilitation, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No